CLINICAL TRIAL: NCT01137825
Title: Carolina Senior: UNC Registry for Older Cancer Patients
Brief Title: Registry of Older Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 0916; P30CA016086 (NIH); CDR0000674085 (Other: PDQ number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Myeloproliferative Disorders; Cognitive/Functional Effects; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Gathering information about older patients with cancer may help the study of cancer in the future.

PURPOSE: This research study is gathering information from older patients with cancer into a registry.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To create a registry (to be called "Carolina Senior") of older patients with an appointment at North Carolina Cancer Hospital.
* To have these patients complete a Geriatric Assessment (GA).

Secondary

* To measure the response rates of GAs of Carolina Senior patients and their satisfaction with a GA by measuring the percentage of patients contacted who consent to complete the GA; the percentage of patients able to complete the self-administered portion of the GA without assistance; the length of time necessary to complete the GA; the variance and number of missing items; the percentage of GAs that contain all 3 of the following items: Timed Up and Go Assessment, Blessed Orientation-Memory-Concentration Test, and healthcare professional-rated Karnofsky performance status; and patient satisfaction with the questionnaire by identifying items that are distressing or too difficult to comprehend.
* To gather information, including patterns of patient care, that would lend support for future research in the 'Carolina Senior' population who receive a confirmed diagnosis of cancer (except for nonmelanoma skin cancer, cervical carcinoma in situ without evidence of disease, or prostatic intraepithelial neoplasia without evidence of prostate cancer).

OUTLINE: Patients complete a geriatric assessment, a multi-dimensional inter-disciplinary patient evaluation that includes an evaluation of a patient's functional status (ability to live independently at home and in the community), co-morbid medical conditions, cognition, psychological status, social functioning and support, medication review, and nutritional status. Patients' medical records are also reviewed. Patients' health status at 1 year is incorporated into the registry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have an appointment at the North Carolina Cancer Hospital and agree to complete the Geriatric Assessment NOTE: Not all patients included in the registry will ultimately be diagnosed with cancer. Patients who complete a GA and are not diagnosed with cancer will remain in the database, but will be categorized into a separate group and will not have their medical records accessed.

PATIENT CHARACTERISTICS:

* Able to read and speak English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Oncology Patients or those with a presumed cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-09; Primary Completion 2030-07-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Creation of a registry of older patients within the University of North Carolina's healthcare system | 4 years
Completion of the Geriatric Assessment (GA) | Upon subject's first visit to the clinic

SECONDARY OUTCOMES:
Information that would lend support for future research | 3 years
  Including patterns of patient care, that would lend support for future research in the 'Carolina Senior' population who receive a confirmed diagnosis of cancer with the exception of:
  * Non-melanoma skin cancer
  * Cervical carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
Response rates of Geriatric Assessments of Carolina Senior patients and their satisfaction with the GA | 2 years
  Done by measuring:
  * Percentage of patients contacted who consent to complete the GA;
  * The percentage of patients able to complete the self-administered portion of the geriatric assessment without assistance;
  * The length of time necessary to complete the geriatric assessment;
  * The variance and number of missing items;
  * The percentage of geriatric assessments that contain all three of the following items: Timed Up and Go Assessment, Blessed Orientation-Memory-Concentration Test, and healthcare professional-rated Karnofsky performance status;

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (7):
- United States (7):
  - Seby B. Jones Cancer Center, Boone, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Pardee Cancer Center, Hendersonville, North Carolina
  - Carteret Health Care Cancer Center, Morehead City, North Carolina
  - Carolina East Radiology, New Bern, North Carolina
  - Rex Healthcare, Raleigh, North Carolina

REFERENCES:
- [Derived] Pergolotti M, Langer MM, Deal AM, Muss HB, Nyrop K, Williams G. Mental status evaluation in older adults with cancer: Development of the Mental Health Index-13. J Geriatr Oncol. 2019 Mar;10(2):241-245. doi: 10.1016/j.jgo.2018.08.009. Epub 2018 Sep 8. PMID 30205939
- [Derived] Guerard EJ, Deal AM, Williams GR, Jolly TA, Nyrop KA, Muss HB. Falls in Older Adults With Cancer: Evaluation by Oncology Providers. J Oncol Pract. 2015 Nov;11(6):470-4. doi: 10.1200/JOP.2014.003517. Epub 2015 Jul 14. PMID 26175532
- See also: web address for Lineberger Comprehensive Cancer Center, UNC — http://unclineberger.org
- See also: web address for the National Cancer Institute (NCI) — http://cancer.gov